CLINICAL TRIAL: NCT03918317
Title: A Study of the Use of AirXpanders AeroForm in Patients Undergoing Post-Mastectomy Radiation Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding unavailable - Company shutting down
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE2119
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- AirXpanders AeroFormtissue expander + Radiation therapy (Experimental): AirXpanders AeroFormtissue expander in participants with breast cancer undergoing post-mastectomy radiation therapy in order to define the toxicity profile and associated subsequent successful surgical reconstruction rate.
  Interventions: Device: AirXpanders AeroFormtissue expander

INTERVENTIONS:
Device: AirXpanders AeroFormtissue expander — The AeroFormdevice will be placed in an immediate fashion at the time of mastectomy in a submuscular, prepectoral or dual-plane approach. The tissue expander will be minimally inflated intraoperatively to minimize dead space and while facilitating tension free closure. Participants will undergo standard postoperative management, and will be given instructions on utilization of the device, including daily expansion until desired volume is reached as determined b surgeon and participant agreement.

SUMMARY:
This study seeks to to determine the efficacy and side effect profile following radiation therapy for participants with the AeroForm device placed. The AeroForm device is FDA approved.

DETAILED DESCRIPTION:
Primary objective:

To assess the proportion of successful initial phase of tissue expander/implant based breast reconstructions (no reconstruction failure or unexpected return to the operating room) following post-mastectomy radiation therapy in participants with AeroFormplaced.

Secondary objectives:

* To evaluate the rate of successful exchange of tissue expander for implant
* To evaluate the rate of reconstruction revisions
* To evaluate CTCAE acute and chronic toxicity rates, infections and cosmetic outcomes
* To evaluate dosimetry to treatment targets as well as organs at risk (heart, lungs) with AeroFormas compared to traditional reconstruction techniques.
* To evaluate time to initiation of chemotherapy and/or radiotherapy.
* To evaluate clinical outcomes-local recurrence, regional recurrence, distant metastases, survival
* To evaluate participant breast reconstruction related QOL with the AirXpander AeroFormdevice

This is a phase II trial evaluating the use of the intervention in participants with breast cancer undergoing post-mastectomy radiation therapy in order to define the toxicity profile and associated subsequent successful surgical reconstruction rate

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically of invasive breast cancer.
* Subjects must be planned for unilateral mastectomy
* Subjects must be planned for reconstruction. Pre-pectoral or sub-pectoral reconstruction allowed. Final reconstruction must be implant
* ECOG Performance status <2
* Subject must have features that will necessitate post-mastectomy radiation therapy:
* Tumors > 5 cm
* Axillary node positive disease (pathologic confirmation)
* Clinical features prior to neoadjuvant chemotherapy to require post-mastectomy radiation therapy
* Recurrent disease without previous radiation
* Clinically node negative participants with positive SLN at surgery
* Internal mammary nodal involvement (clinical assessment)
* Subjects must have no clinical or radiographic evidence of distant metastases (imaging not required unless indicated as part of standard of care)
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving CT simulation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects with metastatic disease
* Subjects receiving any other investigational agents.
* Subjects treated with non-standard radiotherapy (hypofractionation, hyperfractionation, partial breast/axilla)
* Subjects with active infection requiring IV antibiotics
* Subject has a history or current evidence of any condition, therapy, or laboratoryabnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subject has received prior radiation therapy to neck, breast, or chest or other area that will result in overlap.
* Pregnant or breastfeeding women or expecting to conceive children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last day of trial treatment are excluded from this study because of the potential toxicities of radiation therapy. Additionally, because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with AirXpanders, breastfeeding women will be excluded. These potential risks may also apply to other agents used in this study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female gender based on presentation of breast cancer
Enrollment: 0 (Actual)
Dates: Start 2019-07-15 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of successful reconstructions following radiation therapy | up to 6 months following permanent implant placement

SECONDARY OUTCOMES:
Rate of implant success at 6months following replacement. | up to 6 months following permanent implant placement
Rate of reconstruction revisions from Aeroform placement throughout study. | up to 6 months following permanent implant placement
Time to implant exchange from Aeroform placement. | up to 6 months following permanent implant placement
Time to initiation of adjuvant chemotherapy following initial surgery (when applicable). | up to 6 months following permanent implant placement
Time to initiation of radiation therapy following initial surgery | up to 6 months following permanent implant placement
Cosmetic outcomes per the aesthetics scale | up to 6 months following permanent implant placement
  13-question assessment with scores ranging from 13 - 65, higher scores indicating better aesthetics
Quality of life based on the BREAST-Q scales | up to 6 months following permanent implant placement
  Full name BREAST-Q- Reconstruction Module version 2.0, higher is better outcome
Quality of life based on the Breast satisfactions scales | up to 6 months following permanent implant placement
  Full name BREAST-Q- Reconstruction Module version 2.0, higher is better outcome
Number of participants who experience acute toxicity per CTCAE version 4.0 | up to 6 months following permanent implant placement
  See AE/SAE section
Chronic toxicity per CTCAE, Baker scoring | up to 6 months following permanent implant placement
  Full name CTCAE Toxicity/Baker Capsular Contracture, Higher- worse CTCAE and Baker

CONTACTS AND LOCATIONS:
Overall Officials: Chirag Shah, Principal Investigator — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No
Part of sponsored study, not planning to share IPD at this time.